CLINICAL TRIAL: NCT02456259
Title: Postoperative Patency of Internal Jugular Vein After Neck Cannula Insertion in Patients Undergoing Minimally Invasive Cardiac Surgery
Brief Title: Postoperative Patency of Internal Jugular Vein After Neck Cannula Insertion
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Zdenek Turek, MD, Ph.D., University Hospital Hradec Kralove
Other Study IDs: 201504S17P
Record Dates: First submitted 2015-05-24; First posted 2015-05-28 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Surgical Procedure
Keywords: internal jugular vein patency; MICS; neck cannula; Jugular veins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neck cannula group: Patients in this group are indicated for neck cannula insertion due to tzpu of cardiac surgery (MICS)
  Interventions: Procedure: Neck cannula insertion
- Central venous catheter only group: Patients in this group are indicated for central venous catheter insertion only.

INTERVENTIONS:
Procedure: Neck cannula insertion — Neck cannula insertion is necessary for establishing of cardiopulmonary bypass for Minimally Invasive Cardiac Surgery. It is routine procedure for this type of cardiac surgery.
  Groups: Neck cannula group

SUMMARY:
The number of patients undergoing Minimally Invasive Cardiac Surgery (MICS) is increasing each year. MICS procedures on atrioventricular valves are usually performed without conventional sternotomy, an alternative approach is from right anterolateral minithoracotomy. This surgical approach has essential impact both on anesthesia techniques and cardiopulmonary bypass (CPB) settings. Specific anesthesiological procedure is an insertion of neck venous cannula of CPB through the right internal jugular vein into the superior vena cava both for partial and total bypass. The size of neck cannula is between 15 and 21 French depending on the type of surgical procedure and patient's weight. Central venous catheter and eventually sheath are also inserted into the right internal jugular vein. Thus, there is a relevant question regarding postoperative patency of right internal jugular vein in patients undergoing MICS procedures requiring an insertion of neck cannula of CPB. The investigators hypothesize, there is no significant difference in postoperative patency of internal jugular vein assessed by ultrasound in patient undergoing cardiac surgery with and without neck cannula of CPB

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing cardiac surgery

  1. conventional sternotomy without neck cannula as planned operating approach
  2. right minithoracotomy with neck cannula as planned operating approach

Exclusion Criteria:

* Any pathology of right internal jugular vein on preoperative ultrasound (vein not fully compressible, hypoplastic jugular vein, preoperative invasion on right jugular vein)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery both from conventional sternotomy without neck cannula and from right mini thoracothomy reguiring neck cannula insertion into right internal jugular vein.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Postoperative patency of internal jugular vein | 7 days
  Comparison of ultrasound findings on right internal jugular vein preoperatively and 7 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Zdenek Turek, MD, Ph.D., Principal Investigator — University Hospital Hradec Kralove, Dept. of Anesthesiology, Sokolska 581, Hradec Kralove, 50005, Czech Republic
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia

REFERENCES:
- [Background] Vernick WJ, Woo JY. Anesthetic considerations during minimally invasive mitral valve surgery. Semin Cardiothorac Vasc Anesth. 2012 Mar;16(1):11-24. doi: 10.1177/1089253211434591. Epub 2012 Feb 22. PMID 22361820
- [Background] Brass P, Hellmich M, Kolodziej L, Schick G, Smith AF. Ultrasound guidance versus anatomical landmarks for internal jugular vein catheterization. Cochrane Database Syst Rev. 2015 Jan 9;1(1):CD006962. doi: 10.1002/14651858.CD006962.pub2. PMID 25575244